CLINICAL TRIAL: NCT04003181
Title: The Pathogenesis of Chronic Diarrhoea After Treatment for Cancer in Cecum and the Ascending Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other); GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-301-16; 1-16-02-137-17 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2019-04-23; First posted 2019-07-01 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Colon Adenocarcinoma; Diarrhea
Keywords: Bile acid malabsorption; Small intestinal bacterial overgrowth
MeSH Terms: conditions — Colonic Neoplasms; Diarrhea | interventions — Anti-Bacterial Agents; bile acid binding proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive breath test (Active Comparator): Patients with a positive breath test are treated with antibiotics.
  Interventions: Drug: Antibiotics
- Positive SeHCAT scan (Active Comparator): Patients with a positive SeHCAT scan are treated with a bile acid binder.
  Interventions: Drug: Bile Acid Binder
- No intervention (No Intervention): Patients with a normal breath test and a normal SeHCAT scan receive no intervention.

INTERVENTIONS:
Drug: Antibiotics — Ciprofloxacin or Rifaximin for 10 days.
  Arms: Positive breath test
Drug: Bile Acid Binder — Cholestyramine or Colesevelam lifelong.
  Arms: Positive SeHCAT scan

SUMMARY:
Many patients suffer from chronic diarrhoea after surgical treatment for cancer in the right side of the colon.

The investigators' main hypothesis is that colon cancer patients with chronic diarrhoea have a higher risk of bile acid malabsorption compared with colon cancer patients without diarrhoea.

The investigators also expect that a part of the cases of bile acid malabsorption is caused by underlying bacterial overgrowth in the small bowel.

The investigators assume that patients with severe bile acid malabsorption have a lower value of FGF19 in the blood compared to patients with moderate or none bile acid malabsorption.

Furthermore, it is assumed that patients with chronic diarrhoea and documented bile acid malabsorption after surgical treatment for right-sided colon cancer will get improved bowel function when treated with a bile acid binder, or antibiotics in case of bacterial overgrowth.

DETAILED DESCRIPTION:
Patients with chronic diarrhoea after surgical treatment of right-sided colon cancer will be compared to patients without diarrhoea after right-sided colon cancer treatment.

All patients will be asked to answer a short questionnaire regarding bowel function, and they will all have standard blood tests taken to exclude non-cancer related causes of diarrhoea. Besides these standard tests, the value of FGF19 will be measured in a blood sample from the fasting participants. All participants will undergo SeHCAT scan to determine the presence of bile acid malabsorption among right-sided colon cancer patients with and without diarrhoea. In addition, a glucose breath test will be performed to examine, if the patients have small intestinal bacterial overgrowth.

Patients with a positive glucose breath test, and thus bacterial overgrowth, will be treated with antibiotics, followed by another SeHCAT scan, glucose breath test, and measurement of gastrointestinal transit time. In addition, they will be asked to complete the questionnaire regarding bowel function again. All cases with an abnormal SeHCAT scan will be treated with a bile acid binder, and the patients will be asked to complete the questionnaire one more time, and the GITT measurement will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Primary adenocarcinoma in cecum or the ascending colon
* Right-sided hemicolectomy
* Understanding, speaking and reading Danish

Exclusion Criteria:

* Previous major gastrointestinal, urological or gynaecological surgery or oncological treatment
* Radiation therapy
* Recurrence of colon cancer
* Metastasis
* Permanent stoma
* Pregnancy
* Reduced cognitive level that makes it plausible that the patient do not understand the study or is not capable of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Change in SeHCAT retention after 7 days. | The SeHCAT scan consists of a baseline measurement and a measurement after 7 days.
  The diagnosis of bile acid malabsorption in cases vs. controls is determined by a positive SeHCAT scan.
Serum concentration of FGF19 | Through study completion, an average of 1 month.
  The serum value of FGF19 is measured by a blood sample.

SECONDARY OUTCOMES:
Presence of bacteria in the small bowel | Through study completion, an average of 1 month.
  The diagnosis of bacterial overgrowth in the small bowel is determined by a breath test.
Symptom relief after treatment with antibiotics or bile acid binder | After 3 months.
  This will be estimated based on self-reported symptoms: A bowel function questionnaire with 30 questions regarding different aspects of bowel function. The patients should state if they have the symptoms daily, 1-6 times per week, less than once a week, or never.
Quality of life after treatment with antibiotics or bile acid binder | After 3 months.
  This will be estimated based on self-reported symptoms: the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0. A questionnaire with 30 individual questions summing up to form one global health status, five functional subscales, three symptom scales and six single items addressing different aspects of quality of life. The scales range from 0-100 with a higher score representing a higher level of functioning or a higher degree of symptoms, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Laurberg, MD DMSc, Study Chair — Department of Surgery, Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Denmark